CLINICAL TRIAL: NCT04960891
Title: A Cohort IND Expanded Access Program (EAP) for Tebentafusp for Treatment of HLA-A*02:01 Positive Patients With Metastatic Uveal Melanoma
Brief Title: A Cohort IND Expanded Access Program for Supporting Patient Access to Tebentafusp
Acronym: Non Applicable
Status: Available | Type: Expanded Access
Sponsor: Immunocore Ltd (Industry)
Collaborators: Clinigen, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMCgp100-402 EA
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Uveal Melanoma
Keywords: Melanoma; Uveal Cancer; IMCgp100; Immunotherapy; Tebentafusp; Ocular Melanoma; Eye Melanoma; Uveal Melanoma; Gp100; TCR; Bispecific T cell receptor fusion protein; ImmTAC; Immune mobilizing monoclonal T cell receptor against cancer
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — tebentafusp

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Tebentafusp — Concentrate solution for intravenous infusion

SUMMARY:
This Expanded Access Program aims to:

1. Provide access to tebentafusp for mUM patients.
2. Provide access to tebentafusp for patients, who were on the control arm of the randomized controlled Phase II trial (IMCgp100-202) and were unable to crossover during the specified window.
3. Ensure that patients, who are benefiting from tebentafusp treatment while participating in an ongoing Immunocore sponsored clinical study (e.g., IMCgp100-102 or IMCgp100-201), may continue tebentafusp treatment on this Programme once the ongoing trial has met all of its key primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Male or female patients age ≥ 18 years of age at the time of first dose

   Type of Participant and Disease Characteristics
2. Histologically or cytologically confirmed metastatic UM or unresectable UM patients
3. HLA-A*02:01 positive
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

   Informed Consent
5. Ability to provide and understand informed consent prior to procedures [if required]

   Contraception
6. Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control from the trial screening date until 1 week after the final dose of the program intervention; cessation of birth control after this point shall be discussed with a responsible physician.

   1. Pregnant or lactating women are prohibited from enrolling on this program.
   2. Male participants are not allowed to donate sperm from the time of enrolment until 3 months post- administration of program interventions.

Exclusion Criteria:

Disease Under Study and Prior Anticancer Therapy

1. Presence of untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or cord compression. NOTE: Participants with treated CNS lesions may enroll provided all of the following apply:

   1. Treated CNS lesions must be radiographically stable for ≥ 2 weeks after intervention (surgery and/or radiation).
   2. Participants must be neurologically stable off systemic corticosteroids for at least 2 weeks prior to first planned administration of tebentafusp.
2. Receipt of anticancer therapy for the disease under study within the following times prior to the first planned dose of program intervention:

   1. Cellular therapies (e.g., T-cell therapies): 90 days.
   2. Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4)- targeted immunotherapies (e.g., ipilimumab): 28 days
   3. All other immunotherapies, including PD-(L)1-targeted immunotherapies (e.g., atezolizumab, pembrolizumab): 21 days
   4. All other systemic therapies: 14 days
   5. Radiotherapy: 14 days (excepting palliative radiotherapy to a limited field [e.g., for a focally painful tumor mass], which may be administered within 14 days provided there are no ongoing related Grade 2 or higher toxicities)

   Medical Conditions and Concomitant Medications
3. Systemic treatment with steroids or any other immunosuppressive drug use within 2 weeks of the planned first dose of program intervention, with the following exceptions:

   1. Treatment for well-controlled and asymptomatic adrenal insufficiency is permitted, but replacement dosing is limited to prednisone ≤ 12 mg daily or the equivalent.
   2. Local steroid therapies (e.g., optic, ophthalmic, intra- articular, or inhaled medications) are acceptable.
   3. Premedication for allergy to contrast reagent.
   4. Steroids for management of CNS metastases > 2 weeks prior to the planned first dose of program intervention.
4. Any relevant medical condition, which in the opinion of the treating physician, would prevent the participant enrolling into the Program due to concerns related to safety, compliance with procedures, or interpretation of program results.
5. Chronic viral infections as indicated below. NOTE: Testing for hepatitis C virus (HCV) status prior to enrollment is not necessary unless clinically indicated.

   1. Known history of human immunodeficiency virus (HIV) infection.
   2. Known HBV infection, unless on stable anti-viral therapy for > 4 weeks prior to the planned first dose of program intervention and viral load confirmed as undetectable during Screening.
   3. Known HCV infection, unless the participant has received curative treatment and viral load was confirmed as undetectable during Screening.

   Diagnostic Assessments
6. Participant with an out-of-range Screening laboratory values defined as shown below. NOTE: Hematology evaluations must be performed ≥ 7 days from any blood or blood product transfusion and ≥ 14 days from any dose of hematologic growth factor.

   1. Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 30 mL/minute
   2. Total bilirubin > 1.5 × ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin > 1.5 × ULN
   3. Alanine aminotransferase > 5 × ULN
   4. Aspartate aminotransferase > 5 × ULN
   5. Platelet count < 50 × 109/L
   6. Hemoglobin < 8 g/dL
7. Clinically significant cardiac disease or impaired cardiac function, including any of the following:

   1. Congestive heart failure (New York Heart Association Class ≥ 3)
   2. Uncontrolled hypertension defined as systolic blood pressure [BP] > 160 mmHg or diastolic BP > 110 mmHg with the following requirements:

   <!-- -->

   1. If initial measurement is elevated, additional assessments should be taken where each assessment is the mean value of 3 measurements taken at least 5 minutes apart.
   2. Eligibility is based on the average of at least 2 assessments taken at least 1 hour apart.
   3. Acute myocardial infarction or unstable angina pectoris < 6 months prior to the planned first dose of program intervention

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult